CLINICAL TRIAL: NCT06209463
Title: The Effect of Posture, Hand Functions and Sensory Processing Skills on Nutrition in Children With Autism Spectrum Disorder
Brief Title: Posture, Hand Functions and Sensory Processing Skills on Nutrition
Status: Completed | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Collaborators: Istanbul University (Other)
Responsible Party: Principal Investigator, Elif Durgut, ASST.PROF, Bezmialem Vakif University
Other Study IDs: 5325597167
Record Dates: First submitted 2024-01-05; First posted 2024-01-17 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Autism Spectrum Disorder; Autism; Autism, Mild; ASD
Keywords: Autism Spectrum Disorder; posture; sensory processing; hand functions; nutrition
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder; Lymphoma, Follicular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Study group: 40 children with autism underwent postural assessments, including measurement of craniovertebral angle (CVA) for head posture and Pediatric Balance Scale (PBS) for postural control; hand function assessments, including Jebsen Taylor Hand Function Test (JTHFT) for hand skills and Jamar hand dynamometer for hand grip strength; sensory processing assessments using Dunn Sensory Profile; nutrition problem assessments using the Screening Tool of Feeding Problems (STEP) and The Brief Autism Mealtime Behavior Inventory (BAMBI); and evaluation of life quality using the Pediatric Quality of Life Inventory-Parents Form (PedsQL-Parents Form). The Beck Depression Scale (BDI), Beck Anxiety Scale (BAI), and Trait-State Anxiety Scale were used to assess parents depression, anxiety, and anxiety status.
- Control group: 40 typically developing children (control group) underwent postural assessments, including measurement of craniovertebral angle (CVA) for head posture and Pediatric Balance Scale (PBS) for postural control; hand function assessments, including Jebsen Taylor Hand Function Test (JTHFT) for hand skills and Jamar hand dynamometer for hand grip strength; sensory processing assessments using Dunn Sensory Profile; nutrition problem assessments using the Screening Tool of Feeding Problems (STEP) and The Brief Autism Mealtime Behavior Inventory (BAMBI); and evaluation of life quality using the Pediatric Quality of Life Inventory-Parents Form (PedsQL-Parents Form).

SUMMARY:
To examine the effects of posture, hand functions and sensory processing skills on nutrition in children with autism spectrum disorder.

The study aims to include 40 children diagnosed with Autism Spectrum Disorder (ASD), directed from the Department of Child and Adolescent Psychiatry at Istanbul University, along with their parents/caregivers, and 40 healthy children along with their parents/caregivers.

DETAILED DESCRIPTION:
Parents/caregivers of children diagnosed with ASD will be assessed using a demographic information form; sensory processing (Dunn Sensory Profile); nutrition (Screening Tool for Eating Problems (STEP), Brief Autism Mealtime Behavior Inventory (BAMBI)); quality of life (Pediatric Quality of Life Inventory (PedsQL 4.0)); children will undergo assessments for balance (Pediatric Berg Balance Scale); head posture (Craniovertebral angle method), hand functions (Jebsen Taylor Hand Function Test); grip strength (Jamar Hand Dynamometer); and parents' evaluations for depression, anxiety, and stress levels (Beck Depression Inventory, Beck Anxiety Inventory, Spielberger State-Trait Anxiety Inventory).

The assessment duration, including explanations and questionnaires, will take approximately 1 hour.

ELIGIBILITY:
Inclusion Criteria:

* Age between 5-10 years,
* Diagnosis of Autism Spectrum Disorder (ASD),
* Children scoring between 30-36.5 points on the Childhood Autism Rating Scale (CARS),
* Absence of any oral structural disorders,
* Willingness of the parent to voluntarily participate in the study.

Exclusion Criteria:

* Absence of physical, visual, and auditory impairments other than Autism Spectrum Disorder (ASD).
* Presence of any additional neurological, genetic, or metabolic disorders.

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: * Age between 5-10 years,
  * Diagnosis of Autism Spectrum Disorder (ASD),
  * Children scoring between 30-36.5 points on the Childhood Autism Rating Scale (CARS),
  * Absence of any oral structural disorders,
  * Willingness of the parent to voluntarily participate in the study
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2023-11-20 (Actual); Primary Completion 2024-03-20 (Actual); Study Completion 2024-04-04 (Actual)

PRIMARY OUTCOMES:
Craniovertebral angle | 2 weeks
  The craniovertebral angle (CVA) measurement was used to evaluate the head posture of children. The CVA is formed by the angle created by the line connecting the midpoint of the tragus of the ear to the spinous process of C7. A marker was placed on the spinous process of C7 and the tragus. Children were instructed to move their heads up and down, gradually reducing this range of motion. After returning to their natural position, photographs were taken from the right side while looking at a fixed point to ensure correct posture. The photo was then loaded into computer software (MB Ruler 5.0), and the angle was calculated using a triangle ruler between the horizontal line passing through the C7 point and the line extending from the tragus to C7. A decrease in the CVA value (<50 degrees) indicates an increase in anterior head posture. A significant difference was found between the study and control groups in terms of CVA values, in favor of the control group (p<0.05).
Pediatric Balance Scale | 2 weeks
  Pediatric Balance Scale (PBS) was utilized to assess postural control in children. The PBS comprises 14 subdomains, including specific movements such as sitting, standing, turning, and reaching. Each subdomain receives a score between 0 and 4. The maximum achievable score is 56, and a higher score indicates better balance skills.
  A significant difference in PBS scores was found between the study and control groups, favoring the control group (p<0.05).
Jebsen Taylor Hand Function Test | 2 weeks
  Jebsen Taylor Hand Function Test (JTHFT) was used to measure children's hand functions. To conduct the JTHFT, the child was seated in front of the table where the test was administered. The test consists of seven tasks, including writing a 24-word sentence, flipping five cards, picking up small objects, mimicking eating with a teaspoon and five beans, stacking four checkers, picking up and carrying five large empty tin cans, and then picking up and carrying five large full tin cans. A longer duration to perform the tasks clinically indicates a poorer hand skill performance for the child.
  A difference was found between the two groups in terms of all JTHFT subparameter values and handgrip strength values (p<0.05). It was observed that subjects with ASD took longer to perform all JTHFT subtests and had lower handgrip strength values.
Jamar hand dynamometer | 2 weeks
  The measurement of handgrip strength was conducted with the child sitting in a chair, the arm adhered to the body, shoulders in adduction, elbows in 90° flexion, and the forearm and wrist held in a neutral position using a Jamar hydraulic dynamometer with the dominant hand. The child was instructed to grasp the dynamometer firmly and then release it once. A total of 3 measurements were taken with 30-second rest intervals, including 5-second contraction periods. The grip strength values obtained were recorded in kilograms (kg) by taking the average.
  A significant difference was found between the two groups in terms of hand grip strength values (p<0.05). Hand grip strength values were observed to be lower in patients with ASD.
Dunn Sensory Profile | 2 weeks
  Children's sensory processing skills were examined using the Turkish version of the Dunn Sensory Profile. The Dunn Sensory Profile questionnaire is filled out by parents/caregivers to assess the sensory processing skills of children aged 3-10. The questionnaire consists of three main sections. The first part measures children's responses to specific sensory inputs. The second part examines the ability of children to regulate sensory inputs to carry out daily life activities. The third part investigates the behavioral and emotional characteristics that arise when children process sensory information.
  A difference was found between the study and control groups in terms of the Sensory Profile Scale subsection and total scores, in favor of the control group (p<0.05).
Screening Tool of Feeding Problems (STEP) | 2 weeks
  STEP is an instrument that focuses on specific sections by categorizing the occurring feeding problems, highlighting the section it concentrates on. It is a screening tool designed with 23 questions in a Likert-type format. The test contributes to identifying the most commonly observed problem by categorizing observed feeding problems in individuals.
  A difference was found between the study and control groups in favor of the control group in all other STEP subgroup scores except for the 'aspiration risk' score (p<0.05).
The Brief Autism Mealtime Behavior Inventory (BAMBI) | 2 weeks
  BAMBI, developed by Lukens and Lischeid, was used to identify nutritional problems in children [138]. BAMBI consists of 18 items, each presenting 5 different options indicating the frequency of occurrence.An increase in the total score of BAMBI indicates a higher prevalence of specific negative behaviors related to Oral Sensory Processing.
  A difference was found between the study and control groups in terms of BAMBI total score, with the difference favoring the control group (p<0.05).
Pediatric Quality of Life Inventory-Parents Form | 2 weeks
  This scale is a tool used to assess the overall quality of life of children and adolescents aged 2-18. It includes various subdomains such as physical health, emotional function, social function, and school function to measure the quality of life of individuals in different age groups. The higher the total score on Pediatric Quality of Life Inventory-Parents Form , the better the quality of life is perceived to be.
  A difference was found between the study and control groups in terms of Pediatric Quality of Life Inventory-Parents Form subgroups and total scores, favoring the control group (p<0.05). Patients with ASD were observed to have lower Pediatric Quality of Life Inventory-Parents Form scores.
Beck Depression Scale | 2 weeks
  Parents' depression levels were examined using the Beck Depression Inventory (BDI). The BDI is a 21-item questionnaire that assesses the presence and severity of depression. In the scoring system, scores ranging from 0 to 9 indicate minimal depression, 10 to 18 suggest mild depression, 19 to 29 indicate moderate depression, and scores from 30 to 63 indicate severe depression, reflecting the level of depression.
  A difference was found between the study and control groups in terms of BDI scores (p<0.05). It was observed that the parents of ASD patients had higher depression scores.
Beck Anxiety Scale | 2 weeks
  Parents' anxiety levels were assessed using the Beck Anxiety Inventory (BAI). The BAI is a brief 21-item questionnaire that evaluates the severity of anxiety. According to the scoring system, scores ranging from 0 to 9 indicate normal anxiety levels, 10 to 18 suggest mild to moderate anxiety, 19 to 29 indicate moderate to severe anxiety, and scores from 30 to 63 indicate a presence of very severe anxiety.
  A difference was found between the study and control groups in terms of BAI scores (p<0.05). It was observed that the anxiety levels of the parents of the ASD patients were higher.
Trait-State Anxiety Scale | 2 weeks
  To assess the anxiety levels of parents, the State-Trait Anxiety Scale was utilized. This scale is a self-assessment questionnaire consisting of brief statements and provides a four-point Likert-type measurement. Evaluation is based on the responses of parents to questions that ask them to assess each situation. A score of 1 indicates that the specified situation does not reflect themselves at all, while a score of 4 indicates that the situation completely reflects themselves. In the State Anxiety Scale, responses indicate the intensity of emotion, thought, or behavior, while in the Trait Anxiety Scale, they are asked to specify the frequency of these elements. The total score from both inventories can range from 20 to 80. Higher scores represent higher levels of anxiety, while lower scores indicate lower levels of anxiety.
  A difference was found between the study and control groups in terms of State-Trait Anxiety Scale scores (p<0.05).

CONTACTS AND LOCATIONS:
Overall Officials: YAĞMUR AYDOĞAN, Principal Investigator — BEZMIALEM FOUNDATION UNIVERSITY
Locations (2):
- Turkey (Türkiye) (2):
  - Bezmialem Vakıf University, Istanbul, Eyüp
  - Bezmialem Vakıf University, Istanbul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Salahzadeh Z, Maroufi N, Ahmadi A, Behtash H, Razmjoo A, Gohari M, Parnianpour M. Assessment of forward head posture in females: observational and photogrammetry methods. J Back Musculoskelet Rehabil. 2014;27(2):131-9. doi: 10.3233/BMR-130426. PMID 23963268
- [Background] Weinstock-Zlotnick G, Mehta SP. A structured literature synthesis of wrist outcome measures: An evidence-based approach to determine use among common wrist diagnoses. J Hand Ther. 2016 Apr-Jun;29(2):98-110. doi: 10.1016/j.jht.2016.03.001. PMID 27264897
- [Background] Matson JL, Kuhn DE. Identifying feeding problems in mentally retarded persons: development and reliability of the screening tool of feeding problems (STEP). Res Dev Disabil. 2001 Mar-Apr;22(2):165-72. doi: 10.1016/s0891-4222(01)00065-8. PMID 11325163
- [Background] Margari L, Marzulli L, Gabellone A, de Giambattista C. Eating and Mealtime Behaviors in Patients with Autism Spectrum Disorder: Current Perspectives. Neuropsychiatr Dis Treat. 2020 Sep 11;16:2083-2102. doi: 10.2147/NDT.S224779. eCollection 2020. PMID 32982247
- [Background] Posar A, Visconti P. Sensory abnormalities in children with autism spectrum disorder. J Pediatr (Rio J). 2018 Jul-Aug;94(4):342-350. doi: 10.1016/j.jped.2017.08.008. Epub 2017 Nov 4. PMID 29112858
- [Background] Tsujiguchi H, Miyagi S, Nguyen TTT, Hara A, Ono Y, Kambayashi Y, Shimizu Y, Nakamura H, Suzuki K, Suzuki F, Nakamura H. Relationship between Autistic Traits and Nutrient Intake among Japanese Children and Adolescents. Nutrients. 2020 Jul 28;12(8):2258. doi: 10.3390/nu12082258. PMID 32731611
- [Background] Narzisi A, Fabbri-Destro M, Crifaci G, Scatigna S, Maugeri F, Berloffa S, Fantozzi P, Prato A, Muccio R, Valente E, Viglione V, Pecchini E, Pelagatti S, Rizzo R, Milone A, Barone R, Masi G. Sensory Profiles in School-Aged Children with Autism Spectrum Disorder: A Descriptive Study Using the Sensory Processing Measure-2 (SPM-2). J Clin Med. 2022 Mar 17;11(6):1668. doi: 10.3390/jcm11061668. PMID 35329994
- [Background] Matson ML, Matson JL, Beighley JS. Comorbidity of physical and motor problems in children with autism. Res Dev Disabil. 2011 Nov-Dec;32(6):2304-8. doi: 10.1016/j.ridd.2011.07.036. Epub 2011 Sep 3. PMID 21890317
- [Background] Nilsen AKO, Anderssen SA, Johannessen K, Aadland KN, Ylvisaaker E, Loftesnes JM, Aadland E. Bi-directional prospective associations between objectively measured physical activity and fundamental motor skills in children: a two-year follow-up. Int J Behav Nutr Phys Act. 2020 Jan 2;17(1):1. doi: 10.1186/s12966-019-0902-6. PMID 31898547
- [Background] Varni JW, Seid M, Kurtin PS. PedsQL 4.0: reliability and validity of the Pediatric Quality of Life Inventory version 4.0 generic core scales in healthy and patient populations. Med Care. 2001 Aug;39(8):800-12. doi: 10.1097/00005650-200108000-00006. PMID 11468499